CLINICAL TRIAL: NCT07378397
Title: Evaluating Novel OPM-magnetoencephalography in Pre-surgical Mapping for Patients With Epilepsy
Brief Title: OPM MEG in Pre-surgical Mapping for Patients With Epilepsy
Status: Enrolling by invitation | Type: Observational
Sponsor: Aston University (Other)
Collaborators: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: AU-014-2024-CW
Record Dates: First submitted 2026-01-19; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy (Treatment Refractory); Epilepsy in Children; Epilepsy in Youth
Keywords: OPM-MEG; magnetoencephalography
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with epilepsy: Children with refractory epilepsy who are candidates for neurosurgery and have been referred for a clinical MEG scan.

SUMMARY:
Magnetoencephalography, or "MEG", is a brain-scanning method which has been available for many years. It is used in the UK and worldwide to help patients with epilepsy, who need surgery to resolve their seizures. The MEG scan can help inform the surgeon about where to operate, by mapping the abnormal brain activity caused by epilepsy. During a traditional MEG recording, patients sit very still with their head in a rigid helmet which houses many tiny sensors. This can be uncomfortable, and there are additional problems if the patient is a child, because the helmet is often too big. It is not possible to record useful data from the very youngest children with a traditional MEG scanner.

But there is a new generation of MEG systems, called OPM-MEG, which employ lightweight sensors housed in a kind of hat. The hat can be appropriately sized for children, and the patient can move comfortably. The new systems are also more cost-effective to run. It is important to know whether the accepted clinical protocols for using MEG in planning epilepsy surgery can be directly transferred to OPM-MEG. It is also important to understand how the patient experience compares across systems.

In this project, 20 volunteer patients will be recruited from among those children already having routine pre-surgical MEG recordings Aston University. They will be invited to participate in an OPM-MEG recording in the same facility at Aston University, so that data from the new OPM-MEG device can be compared with the data from the old MEG scanner. Data analysis pipelines will be streamlined, and the accuracy of the results compared to determine whether the improved sensor arrangement for children in the OPM-MEG system leads to better localisation of epileptiform activity.

DETAILED DESCRIPTION:
1. BACKGROUND

   Magnetoencephalography (MEG) is a non-invasive brain imaging technique which offers unique, non-redundant clinical information in the planning of surgery for patients with epilepsy. The MEG data are used to localise the inter-ictal activity that in turn can help formulate hypotheses on the localisation of the seizure onset zone. Better outcomes are associated with earlier surgery (i.e., when a child is younger), and with greater preservation of functional tissue. Aston IHN has been offering a MEG service to children and adults awaiting neurosurgery for two decades.

   MEG works by measuring the magnetic fields that indicate the electrical signatures of neural populations acting in synchrony. The established MEG technology relies on cryogenic cooling of the sensors to obtain very high sensitivity, and therefore traditional MEG devices are bulky with a rigid helmet, and also expensive to run. The patient is required to remain very still during the recording, which can be uncomfortable especially for children. Furthermore, the majority of MEG systems worldwide are designed for adult-sized heads and provide poor signal to noise ratios in younger patients.

   There is a new generation of MEG systems called OPM-MEG systems. With a different sensor design, these "wearable" devices operate at or near room temperature and make use of a lightweight helmet or hat that can allow the patient to move during recordings and can be sized appropriately for any age. In theory, OPM-MEG promises better data quality, because sensors are closer to the head (increasing signal), and may improve the efficacy of MEG as a pre-surgical diagnostic tool by increasing spatial resolution and inter ictal discharge detection.

   The aim of this research is to enable the direct comparison of OPM-MEG with traditional (cryogenic) MEG, so that it can be determined whether the new OPM-MEG technology offers the same benefits to patients. Specifically the aim is to record data on both devices, for a small series of 20 cases, and to develop parallel analysis routines to compare the accuracy of the results obtained from each device.
2. RATIONALE OPM-MEG devices employ different sensor technology from traditional cryogenic MEG systems; also, the sensors are also placed closer to the scalp, and in a less dense configuration. There are additional variations in sensor properties such as signal to noise ratio which when coupled with variations in sensor placement can alter the detectability of brain signals. Furthermore, interpretation of MEG data relies on analysis software pipelines, the vast majority of which have been developed for cryogenic MEG.

Before OPM-MEG can be fully validated for clinical work with patients, it is necessary to establish the equivalent data recording and data analysis pipelines, that enable direct comparison between the outputs of each measurement technique. Specifically, for pre-surgical MEG measurements in patients with epilepsy, it is important to know whether OPM-MEG can replicate or improve upon the spatial accuracy and signal sensitivity of cryogenic MEG in identifying inter-ictal abnormalities in brain data that can help identify the epileptogenic source.

Theoretical studies do suggest that OPM-MEG should offer sufficient sensitivity, but there is a lack of available patient data to enable the development of realistic data processing pipelines for a systematic comparison between the two kinds of system. This study therefore aims to collect a case-series of datasets where the same patient has participated in a MEG recording on both a traditional cryogenic MEG system and a novel OPM MEG system. These data will be used to refine data processing pipelines, to explore the patient experience, and to perform an initial comparative study between the two systems.

This work is worthwhile to patients, because if OPM-MEG is found to be at least equivalent to traditional cryogenic MEG it offers, firstly a much more ergonomic, comfortable recording environment where patients can move instead of being in a restricted position. Secondly, the helmet housing the sensors can easily be adjusted to fit children of all ages, meaning that MEG can contribute to pre-surgical evaluations in the youngest patients who currently don't fit in a traditional system. Finally, OPM-MEG systems, not requiring cryogenic cooling, are much cheaper to run than the traditional MEG systems and therefore potentially more cost-effective. In summary, OPM-MEG has the potential to benefit much greater numbers of patients than traditional cryogenic MEG.

ELIGIBILITY:
All patients referred to the Aston IHN MEG service from Birmingham Children's Hospital Children's Epilepsy Surgery Service, who are between the ages of 6 and 15, are eligible to take part in the study, until 20 patients have completed the study.

Inclusion criteria for patients

* Patients who are capable of giving informed assent, and have a person with parental responsibility capable of giving informed consent on their behalf.
* Male or female.
* Patients between the age of 6-15 years
* Patients and caregivers with English language skills that enable informed assent/consent.

Exclusion criteria for patients

• Patients, or parent or caregiver, who do not assent or consent to participate in the research either on that day or later.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population is all children who are in the care of Birmingham Children's Hospital Epilepsy Surgery Service, who have been referred to Aston University for a clinical MEG scan as candidates for neurosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Comparative localisations of epileptiform activity | Within 3 months of referral
  Interictal epileptiform activity recorded in the OPM-MEG data will be localised with standard techniques, and resulting brain activity maps compared with those obtained in cryogenic MEG data that is shared into the study.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline WITTON, PhD, Principal Investigator — Aston University
Locations (1):
- Aston University, Birmingham, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is essentially a qualitative proof of concept study and data may not be of the required quality for sharing.